CLINICAL TRIAL: NCT03778372
Title: Methadone for Emergence Delirium in Children Undergoing Outpatient Strabismus Surgery
Status: Completed | Type: Observational
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Khaled Dajani, Assistant Professor, Ochsner Health System
Other Study IDs: Pro00014855
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Emergence Delirium; Strabismus
MeSH Terms: conditions — Emergence Delirium; Strabismus | interventions — Methadone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- study: pediatric patients undergoing outpatient strabismus surgery, and receiving methadone
  Interventions: Drug: Methadone
- control: pediatric patients undergoing outpatient strabismus surgery, and not receiving methadone

INTERVENTIONS:
Drug: Methadone — see desc above
  Groups: study

SUMMARY:
Strabismus surgery for children is a very common procedure, with a high incidence of emergence delirium in the recovery room. Pain is often implicated in delirium. The primary aim of this study is to determine whether a single, intraoperative dose of methadone for outpatient ambulatory pediatric strabismus surgery reduces postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II children undergoing outpatient strabismus surgery

Exclusion Criteria:

* anything not meeting the above

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy children, aged 0-18 years, undergoing outpatient strabismus surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2020-12-13 (Actual)

PRIMARY OUTCOMES:
Pediatric Anesthesia Emergence Delirium scale scores | measured every 10 minutes in the recovery room, until patient is discharged, up to 6 hours.
  A low total score would indicate less emergence delirium

SECONDARY OUTCOMES:
wong-baker or numeric pain scores, depending on age | measured every 10 minutes in the recovery room, until patient is discharged, up to 6 hours.
  A low total score would indicate less pain
discharge time | 24 hours
  time the patient is actually discharged from recovery room

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Main Campus, Jefferson, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Komen H, Brunt LM, Deych E, Blood J, Kharasch ED. Intraoperative Methadone in Same-Day Ambulatory Surgery: A Randomized, Double-Blinded, Dose-Finding Pilot Study. Anesth Analg. 2019 Apr;128(4):802-810. doi: 10.1213/ANE.0000000000003464. PMID 29847382
- [Background] Ward RM, Drover DR, Hammer GB, Stemland CJ, Kern S, Tristani-Firouzi M, Lugo RA, Satterfield K, Anderson BJ. The pharmacokinetics of methadone and its metabolites in neonates, infants, and children. Paediatr Anaesth. 2014 Jun;24(6):591-601. doi: 10.1111/pan.12385. Epub 2014 Mar 26. PMID 24666686